CLINICAL TRIAL: NCT01702246
Title: Phase 2 Study of Simvastatin Treatment Effects on Vaso-occlusive Pain in Sickle Cell Disease
Brief Title: Effect of Simvastatin Treatment on Vaso-occlusive Pain in Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Carolyn Hoppe, Associate Hematologist-Oncologist, UCSF Benioff Children's Hospital Oakland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDCF-ICRA-2011
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; statins; vaso-occlusive pain; inflammation; biomarkers
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- simvastatin (Experimental): Simvastatin (Zocor), 40mg tablet, 40mg orally once daily, for 3 months
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 40 mg, orally, once daily for 3 months
  Other Names: Zocor

SUMMARY:
The purpose of this study is to determine whether simvastatin is effective in reducing the frequency and intensity of vaso-occlusive pain episodes in patients with sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is characterized by recurrent vaso-occlusive episodes and a chronic inflammatory state leading to progressive multi-organ injury. The pathophysiology of SCD is related to endothelial dysfunction driven largely by impaired nitric oxide (NO) homeostasis and chronic inflammation. Through multiple mechanisms, including upregulation of NO, statins have been shown to confer protection from endothelial injury, independent of their cholesterol-lowering properties.

By inhibiting inflammation and several common pathways leading to vascular damage,simvastatin may help prevent the acute and chronic complications of SCD. The objective of this study is to determine whether our preliminary results showing simvastatin-associated reductions in plasma markers of vascular injury will translate into a reduction in vaso-occlusive pain episodes in patients with SCD. A web-based, smartphone-accessible electronic pain diary will be used to monitor frequency and intensity of vaso-occlusive pain in SCD patients treated with a single daily dose of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease (HbSS or S/β0 thalassemia)
* ≥ 3 vaso-occlusive pain episodes in the year prior to enrollment
* Age ≥ 10 years
* Weight > 30 kg

Exclusion Criteria:

* Creatine kinase (CK) > UNL
* Total cholesterol < 90 mg/dL, or triglycerides <30mg/dL
* Renal dysfunction (Creatinine > 1.5-fold UNL)
* Hepatic dysfunction (ALT > 2-fold UNL)
* Treatment with drugs having known metabolic interactions with statins within the past 30 days
* Vaso-occlusive pain requiring hospitalization within past 30 days
* Red blood cell transfusion within the past 30 days
* Pregnancy/lactation
* Musculoskeletal disorder associated with an elevated CK level
* Past or present history of substance abuse (alcohol, cocaine, amphetamines, heroin)
* Chronic pain caused by avascular necrosis of the bone (AVN) or leg ulcers, and pain due to trauma or causes other than SCD.
* Major cognitive or neurological impairments that may hamper the ability to use the smartphone or complete the electronic pain diary in this study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Hoppe, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital and Research Center Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No
publication

REFERENCES:
- [Background] Hoppe C, Kuypers F, Larkin S, Hagar W, Vichinsky E, Styles L. A pilot study of the short-term use of simvastatin in sickle cell disease: effects on markers of vascular dysfunction. Br J Haematol. 2011 Jun;153(5):655-63. doi: 10.1111/j.1365-2141.2010.08480.x. Epub 2011 Apr 8. PMID 21477202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin
Started | 24
Completed | 19
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Simvastatin
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Receiving hydroxyurea (HU) therapy [Number; unit: participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Vaso-occlusive Pain Events, Before and After Treatment With Simvastatin
Description: The effect of simvastatin treatment will be assessed by measuring the difference from baseline in the mean frequency (and intensity) of vaso-occlusive pain events, after treatment with simvastatin. Pain rate (proportion of pain days) was defined as the number of days reported with sickle cell disease-related pain divided by the number of daily pain diaries completed.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: proportion of pain days
Groups:
- Baseline: prior to treatment with simvastatin
- Simvastatin: after treatment with simvastatin: 40 mg, orally, once daily for 3 months
Arm/Group | Baseline | Simvastatin
Number analyzed (Participants) | 19 | 19
proportion of pain days | 0.2365 (0.21) | 0.1311 (0.15)
Statistical Analysis 1: Comparison: Baseline vs Simvastatin; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney) — Wilcoxon matched pairs signed rank test

2. Secondary Outcome: Change in Plasma High Sensitivity C-reactive Protein
Description: Mean difference in plasma high sensitivity C-reactive protein level, before and after treatment with simvastatin
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Baseline | Simvastatin
Number analyzed (Participants) | 19 | 19
mg/mL | 7.2 (11) | 2.989 (4.169)
Statistical Analysis 1: Comparison: Baseline vs Simvastatin; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Total Cholesterol Level After Treatment With Simvastatin
Time Frame: Baseline and 3 months
Population: change in baseline cholesterol level from baseline, after treatment with simvastatin
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Baseline Cholesterol: mean cholesterol level (mmol/L) prior to treatment with simvastatin
- Simvastatin Treatment: after treatment with simvastatin: 40 mg, orally, once daily for 3 months
Arm/Group | Baseline Cholesterol | Simvastatin Treatment
Number analyzed (Participants) | 19 | 19
mmol/L | 124 (27) | 101 (17)
Statistical Analysis 1: Comparison: Baseline Cholesterol vs Simvastatin Treatment; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Safety data were collected on each participant during the treatment period (3 months) and at 1 month follow up
Arm/Group | Simvastatin
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin (N=19)
sickle cell vaso-occlusive pain crisis (Blood and lymphatic system disorders) | 4 — Four participants were hospitalized for sickle cell related vaso-occlusive pain crisis (expected SAE)
hyperhemolysis (Blood and lymphatic system disorders) | 1 — One participant was hospitalized for sickle cell related hyperhemolytic event (unrelated to study drug)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=19)
facial rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No